CLINICAL TRIAL: NCT02283684
Title: Green Light Laser (XPS) Photoselective Vaporization of the Prostate (PVP) Versus Bipolar Transurethral Vaporization (B.TUVP) of the Prostate for Treatment of Small to Moderate Sized Benign Prostate Hyperplasia: A Randomized Study
Brief Title: GreenLight Laser Photoselective Vaporization of the Prostate vs Bipolar Transurethral Vaporization of the Prostate; RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Lecturer of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mans-2014-03
Record Dates: First submitted 2014-11-02; First posted 2014-11-05 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: LASER; PROSTATE; BIPOLAR; HYPERPLASIA; VAPORIZATION
MeSH Terms: conditions — Prostatic Hyperplasia; Hyperplasia | interventions — Photoelectron Spectroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Greenlight laser PVP (Active Comparator): Greenlight (532-nm) laser Photoselective vaporization of the prostate using (XPS) 180W system
  Interventions: Procedure: Greenlight laser PVP
- Bipolar TUVP (Active Comparator): Bipolar transurethral vaporization of the prostate using bipolar system
  Interventions: Procedure: Bipolar TUVP

INTERVENTIONS:
Procedure: Greenlight laser PVP — Vaporization of the prostate adenoma using 532nm laser with 180W XPS system using Moxy fiber
  Other Names: Greenlight (532-nm) laser PVP using (XPS) 180W system
  Arms: Greenlight laser PVP
Procedure: Bipolar TUVP — Bipolar energy is used for generation of plasma that ends up by vaporization of the prostate adenoma
  Arms: Bipolar TUVP

SUMMARY:
With a growing body of knowledge on the promising advancements and recent clinical data of the third generations of the Greenlight PVP/XPS, it seems to be a real contender in the world of MIS. Contenders of Greenlight laser technology includes bipolar as well as Holmium laser technology.

In this study the investigators planned to test the Greenlight (532-nm) laser PVP using (XPS) 180W system compared to bipolar electro-vaporization, in reduction of LUTS secondary to small to moderate sized BPH in a prospective randomized trial.

DETAILED DESCRIPTION:
Patients with LUTS due to BPH seen through the outpatient prostate clinic in the Mansoura UNC were assessed to evaluate if the patient is eligible to the study inclusion criteria. Patients who are meeting these criteria were asked to participate in this randomized comparative study and were provided with an informed consent form. Study participants were enrolled and randomized, and the appropriate scheduled procedures were performed.

Preoperatively, all patients were thoroughly evaluated by medical history and physical exam, digital rectal exam (DRE), prostate specific antigen (PSA), urinalysis and urine culture, international index of prostate symptom score (IPSS), Quality of Life (QOL), transrectal ultrasound (TRUS) measurement of prostatic volume and biopsy whenever indicated, measurement of post-void residual assessment (PVR), and maximum urinary flow rate (Qmax). Preoperative flexible urethrocystoscopy was done when hematuria was the presenting symptom.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age ≥50 years
2. LUTS secondary to BOO due to BPH who failed medical treatment
3. International prostate symptom scores (IPSS) >15 and bother score (QOL) ≥ 3 (according to IPSS question 8)
4. Peak urinary flow rate (Qmax) <15 ml/sec with at least 125 ml voided volume or Patients with acute urine retention secondary to BPH who failed trial of voiding on medical treatment.
5. ASA (American society of anaesthesiologists) score ≤3.
6. TRUS prostate size (from 30 to 80ml)

Exclusion Criteria:

1. Patient with neurological disorder which might affect bladder function as cerebrovascular stroke, Parkinson disease
2. Active urinary tract infection,
3. Presence of active bladder cancer (within the last 2 years)
4. Known prostate cancer patients will be excluded preoperatively on the basis of digital rectal examination, prostate specific antigen level, and TRUS imaging followed by prostate biopsies if necessary.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
IPSS change | two years
  change in the symptoms score over two years post procedure

SECONDARY OUTCOMES:
Reoperation rate | 4 years
  need for reintervention post procedure
Q.max | 2 years
  maximal urine flow rate
biopsy | one month
  clinicopathological outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt